CLINICAL TRIAL: NCT03200795
Title: Effect of Rebound Exercises and Circuit Training on Musculoskeletal Pain, Selected Biochemical and Psychosocial Parameters Among Individuals With Type 2 Diabetics
Brief Title: Effect of Different Exercises on Musculoskeletal Pain,Glucose Level and Quality of Life Among Patients With Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of KwaZulu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 4198
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2017-06

CONDITIONS: Diabetes
Keywords: Diabetes; Musculoskelatal pain; Rebound exercises; Depression; Glucose; Quality of life
MeSH Terms: conditions — Diabetes Mellitus; Depression | interventions — Circuit-Based Exercise

STUDY DESIGN:
Intervention Model Description: There will be 3 group, the rebound exercise group, circuit training group and the control group. The rebound exercises group will received rebound exercise therapy while circuit training will received circuit exercises that comprises progressive resistance exercise and aerobic exercises, while control group will be treated based on the guideline of the management of diabetes by international diabetes federation. Also the two exercise group will received their routine care plus exercises.
Who Masked: Participant
Masking Description: To eliminate bias, the assessment of outcome will be performed by (experienced) blinded assessors, who will be blinded to the type of intervention as well as the intervention groups of the participants. Participants will also be instructed not to disclose their individual intervention groups to the assessors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rebound exercise group (Experimental): Participants randomized to this group will be instructed on the proper techniques of the desired movements (hopping) on the rebounder.
  Interventions: Other: Rebound exercise
- Circuit training group (Experimental): The circuit training for the participants in this group will be designed for each participant. Training will take place 3 times a week for 8 weeks. The participants will undergo 10 minutes warm up before and 10 minutes cool down after the training. Resistance exercises will be performed on weight machines. Throughout the resistance training program, participants will be alternating between the bench press, seated row, lateral pull down, biceps forward, front thigh, back thigh, leg press and rowing.
  Interventions: Other: Circuit training exercise

INTERVENTIONS:
Other: Rebound exercise — Each participant will undergo 3 sessions a week for 8 weeks with each session lasting 20 minutes. Bouncing frequency will be determined by signals from an metronom and will be set at between 90 and 120 bounces per minute. Heart rate training zone will be maintained, during the exercise, at moderate intensity of 40-60% and will be calculated using the Karvonen formula ([Heart rate reserve x training percentage] + resting heart rate)(Nuhu & Maharaj, 2017).
  The exercise will involve bouncing on the center portion of the mini trampoline (Portable 2013 Model Half-Fold Cellerciser with feet slightly apart and knees in full extension. Each foot strike equaled one step or bounce with step height, this will be defined as the distance between the foot at maximum height of jump and the bed of the center of the trampoline ranging between 10 and 15 cm (Nuhu & Maharaj, 2017).
  Arms: Rebound exercise group
Other: Circuit training exercise — Participants will be instructed to exhale while lifting a weight and inhale while lowering it, to minimize blood pressure excursions, and to rest for 2 to 3 minutes between sets. Participants will perform 1 set per resistance exercise three time weekly for the first 2 weeks and 4 sets of each resistance exercise three time weekly during weeks 3 and 4. Resistance will be increase by 5 to 10 kg when the participant could perform more than 15 repetitions while maintaining proper form.
  All aerobic activities of the circuit training will be performed on a cycle ergometer or treadmill. Participants are free to vary the machine used from one visit to the next. Exercise intensity will be standardized by using heart rate monitors (Polar Electro Oy) that will display the participant's heart rate and emitted a warning signal when the heart rate was outside the prescribed training zone, thus guiding the participant in adjusting the workload up or down to achieve the desired intensity.
  Arms: Circuit training group

SUMMARY:
Background. Diabetes is a global epidemic disease. The prevalence of diabetes for all age groups worldwide was estimated to be 2.8% in 2000 and is predicted to affect 4.4% by 2030. The global prevalence of diabetics is currently estimated to be 285 million and projection rates are expected to rise to over 438 million by the year 2030, with Asians suffering the bulk of the total diabetes epidemic.

The incidence of chronic diseases of lifestyle such as Type 2 Diabetes Mellitus (DM) is on the increase amongst the South African population. Due to the numerous factors such as lack of education, inaccessibility of healthcare facilities and/or poor socio-economic background, diabetes mellitus often goes undetected in rural areas, resulting in an increase in musculoskeletal complication and other diabetes mellitus complications. Inability to control blood sugar may induce serious complications such as renal disease, peripheral neuropathy, retinopathy, and vascular events. Due to its multi-systemic nature, diabetes will lead to the development of additional manifestations such as musculoskeletal complications, reduces respiratory capacity, depression and poor quality of life.

Studies have shown that both exercises and pharmacotherapy can decreases depression and improved glycemic control and overall quality of life of persons with diabetes. Thus, in addition improve the quality of life and substantial financial savings and improved medical care of these individuals.

Hypothesis

1. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients at the baseline and at the end of 8 weeks of rebound exercises.
2. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients at the baseline and at the end of 8 weeks of circuit resistance training.
3. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients at the baseline and at the end of 8 weeks of routine care.
4. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients between the rebound exercises group, circuit training and routine care at the baseline.
5. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients between the rebound exercises group, circuit training and routine care at the end of 8 week of the programme.

Summary of the proposed research methodology. The participants will be randomised into three groups. The first group will be engaged in rebound exercise, the second group will be engaged in circuit training while the third group will continue with their normal care of medication. But before the commencement of the study, pilot study will be conducted on normal subjects. Measurement will be carried out at the baseline, four weeks and at the end of the programme, 'The following parameters will be measured. Pain level, blood glycemic level of each participant, cholesterol level, depression and quality of life.

DETAILED DESCRIPTION:
Background Diabetes is a global epidemic disease. The prevalence of diabetes for all age groups worldwide was estimated to be 2.8% in 2000 and is predicted to affect 4.4% by 2030. The global prevalence of diabetics is currently estimated to be 285 million and projection rates are expected to rise to over 438 million by the year 2030, with Asians suffering the bulk of the total diabetes epidemic.

The incidence of chronic diseases of lifestyle such as Type 2 Diabetes Mellitus (DM) is on the increase amongst the South African population. Due to the numerous factors such as lack of education, inaccessibility of healthcare facilities and/or poor socio-economic background, diabetes mellitus often goes undetected in rural areas, resulting in an increase in musculoskeletal complication and other diabetes mellitus complications resulting in increased in diabetes and its complications. Inability to control blood sugar may induce serious complications such as renal disease, peripheral neuropathy, retinopathy, and vascular events. Due to its multi-systemic nature, diabetes will lead to the development of additional manifestations such as musculoskeletal complications, reduces respiratory capacity, depression and poor quality of life.

Musculoskeletal (MSK) complications of diabetes mellitus (DM) are the most common endocrine arthropathies. These have been generally under-recognized and poorly treated compared with other complications, such as neuropathy, retinopathy, and nephropathy. These manifestations, which are some of the causes of chronic disability. This involve not only the joints, but also the bones and the soft tissues. In 2004, the National Health Interview Survey determined that 58% of diabetic patients would have functional disability. The percentage of diabetic patients with functional disability will increase as the number of diabetic patients increases, and hence constitute a major public health problem. Recent data show that the prevalence of MSK manifestations in the hands and shoulders in patients with type 1 or type 2 diabetes is 30%. These manifestations are closely linked to age, prolonged disease duration, and vascular complications in the form of retinopathy.

Depression have been associated with diabetes these depressive symptoms are more likely to persist among persons with multiple diabetic-related complications like musculoskeletal disorders. Studies have shown that both exercises and pharmacotherapy can decreases depression and improved glycemic control and overall quality of life of persons with diabetes. Thus, in addition improve the quality of life and substantial financial savings and improved medical care of these individuals.

Musculoskeletal disorders and disability are very common in diabetes and are associated with worse glycemic control and more complications. Assessment of musculoskeletal disorders among diabetes should include an estimate of cholesterol, glycemic control, pain, respiratory parameters and quality of life. People with diabetes are twice at risk of suffering from premorbid depression as the general population. The coexistence of depression in people with diabetes catalyses serious disease comorbidities, MSK complications, decreased respiratory capacity, poor glycemic control which may lead to hyperlipidemia and poor quality of life and escalated healthcare expenditures.

Rebound exercise is the therapeutic movement on the mini trampoline, it moves all parts of the body at once so it is also call a cellular exercise. It may be superior to any other exercises because is not only uses gravity but also two other forces, acceleration and deceleration at the top of the bounce you experience weightlessness, and at the bottom your weight doubles pulling into the centre of the rebounder. While circuit training is combination of strength training and aerobic exercises. Strengthening training exercises is a resistance exercise that helps to keep the muscle flexible and strong and also strengthens the bones. Aerobic exercise on the other hand is more vigorous exercises that increase oxygen consumption, increase in oxygen consumption helps to burn more calories, stimulate immune response and cardiovascular health.

Appropriate level of exercises such as rebound exercises can aid the management of type 2 diabetes and is likely to improve musculoskeletal Pain and depression. Circuit resistance training has recently been documented to be a safe in the management of type 2 diabetics; however, its effects on MSK pain and depression have not been assessed. Previous studies that assessed resistance exercise with combined resistance and aerobic exercise sessions, showed significant reductions in HbA1c. In contrast, other researchers did not observe any favourable changes in fasting glucose or HbA1c in patients with type 2 diabetes and did not assess its effect on MSK pain, respiratory parameters, depression and quality of life.

Rehabilitation can assist to retrain physical and functional abilities as well as psychological emotions. Therefore, comprehensive rehabilitation to diabetes patients that encompasses exercises like rebound and circuit training may improved glycemic functions and reduces musculoskeletal functions and is very important to mitigate the negative impact has on a person with diabetes.

Exercise has been documented as effective in the management of MSK pain, however there is no consensus regarding the type of exercises that improve MSK pain, and if exercise is effective in reducing depression and improvement in respiratory function among individuals with type 2 diabetes has not been documented.

STATEMENT OF PROBLEMS Diabetes mellitus (DM) is a multi-system disease characterized by persistent hyperglycemia and has both acute and chronic biochemical and anatomical sequelae. Type 2 DM represents approximately 90% of all cases of diabetes.

Previous studies have assessed the effect of resistance exercise with combined resistance and aerobic exercise sessions on type 2 DM and showed significant reductions. However, Balagopal, Kamalamma, Patel, & Misra, 2008 did not observe any favorable changes in fasting glucose or HbA1c in patients with type 2 diabetes. Therefore, there is no consensus on the effect of circuit resistance training (CRT) in type 2 diabetes. To the best of my knowledge, no clinical trial has been conducted that compares the effect of rebound exercises and circuit training on MSK pain, respiratory parameters and psychosocial variables among patients with type 2 diabetes.

Cochrane review recommended that the features studies for the effect of exercises in the management of type 2 diabetes should focus on quality of life, depression and effect on some complication like musculoskeletal pain or disorders and cardiorespiratory fitness.

In African countries, there is a paucity of reports that describe MSK disabilities in diabetic patients. To best of my knowledge no previous studies had been conducted to assess the effect of any treatment of MSK manifestations in diabetic patients or to evaluate the predisposing factors. This study is therefore proposed to determine the effect of rebound exercises and circuit training on musculoskeletal pain, as well as selected biochemical and psychosocial factors among individuals with type 2 diabetes.

RESARCH QUESTION 5. What is the effect of 8 weeks of rebound exercises training on glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients? 6. What is the effect of 8 weeks of circuit resistance training on glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients? 7. What is the effect of 8 weeks of routine care (control group) of medication and counselling as recommended by international diabetic federation (IDF) on glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients? 8. Is there any significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients in the control group, the rebound exercises group and the circuit resistance training group? AIMS AND OBJECTIVES The major aim of this research is to investigate the effect of rebound exercises and circuit training and compare them to the routine care of type 2 diabetic patient Specific objectives of the study

1. To determine the effect of rebound exercises on glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients.
2. To determine the effect of circuit resistance training on glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients
3. To determine the effect of routine care (control group) on glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients.
4. To compare the effect of circuit training, rebound exercises and routine care on glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients
5. Hypothesis
6. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients at the baseline and at the end of 8 weeks of rebound exercises.
7. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients at the baseline and at the end of 8 weeks of circuit resistance training.
8. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients at the baseline and at the end of 8 weeks of routine care.
9. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients between the rebound exercises group, circuit training and routine care at the baseline.
10. There will be no statistical significant difference in glycemic control, cholesterol level, respiratory parameters, pain scores, depression and quality of life among type 2 diabetes patients between the rebound exercises group, circuit training and routine care at the end of 8 week of the programme.

Significance of the study

The outcome of this study is expected to:

4. Provide additional strategy in glycemic control, cholesterol level, respiratory parameters, musculoskeletal pain, depression and quality of life among type 2 diabetes patients by promoting the use of exercises.

5. Show which exercise is the most effective in glycemic control, cholesterol level, respiratory parameters, musculoskeletal pain, depression and quality of life among patients with type 2 diabetes.

6. Give insight into the nature of musculoskeletal pain among type 2 diabetes patients.

Methods Ethical approval will be sought and obtained from University of KwaZulu-Natal Biomedical research ethics committee, before the commencement of the study. Assessment of participants will be conducted at three stages baseline, four week of intervention and at the end of eight week of interventions. To ensure a comprehensive assessment, we chose a battery of measures covering the WHO-ICF model. We selected certain tools to cover the three key domains proposed by the ICF: body structures and function, activity and participation. At baseline, participants will be assessed for socio-demographic characteristics which will include personal demographic information and diabetes specific information. The personal demographic information will include age, sex, height, weight, marital status, educational qualification, employment. The diabetes specific information will include, type of diabetes. At the baseline, the outcome measures to be used for these assessments are presented in the measurement section.

Pilot study Pilot study will be conducted before the commencement of the study, the pilot study will enable the researcher and the research assistant to familiarized them self with the protocol of the intervention. The pilot study will involve two group the rebound exercises group and the circuit training group, each group will have at least 10 participants and they will be recruited from the gymnasium of the department of Biokinetic and physiotherapy School of Health sciences, College of Health Sciences, University of KwaZulu-Natal.

Participants The participants for the study will include patients diagnosed with type 2 diabetes, who will be screened for musculoskeletal pain using the Nordic musculoskeletal symptoms questionnaire. They will also be screened for depression using the Beck Depression Inventory (BDI). Only subjects with musculoskeletal symptoms and depression will be included in the study. The consent of the subjects will be sought before they participate in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with diagnosis of type 2 diabetes for at least 4 years on oral hypoglycemic control
2. Age between 20 to 55 years
3. Musculoskeletal affectation and depression,
4. Consent to participate in the study.

Exclusion Criteria:

1. Subjects who are involved in sporting activities
2. Those whose musculoskeletal problems are severe and may prevent them from performing some of the exercises.
3. Individuals with hypertension
4. Coronary artery disease
5. Myocardial infarction
6. Cardiac or abdominal surgery
7. Previous 6 months, history of fractures of the spine, hip, knee and ankle joints
8. Lower limb weakness and deformities with loss of protective sensation in the feet.
9. Pregnancy or lactation
10. Use of insulin
11. Presence of retinopathy,
12. Nephropathy
13. Subjects who do not consent to participate.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2018-11-20 (Estimated); Study Completion 2019-02-20 (Estimated)

PRIMARY OUTCOMES:
Pain Change is being assessed | Baseline and at the end of eight week of the study
  Musculoskeletal pain will be assess, using visual analog scale (VAS)
Blood glucose level Change is being assessed | Baseline and at the end of eight week of the study
  The sugar level will be measure using accutrend plus
Cholesterol level Change is being assessed | Baseline and at the end of eight week of the study
  The cholesterol level will be measure using accutrend pus

SECONDARY OUTCOMES:
Depression Change is being assessed | Baseline and at the end of the eight week of the study
  The depression will be measure using Beck depression inventory
Quality of life Change is being assessed | Baseline and at the end of the eight week of the study
  The quality of life will be measure using the short form health survey questionnaire (SF-36)

CONTACTS AND LOCATIONS:
Locations (1):
- Aminu Kano Teaching Hospital, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Misra A, Alappan NK, Vikram NK, Goel K, Gupta N, Mittal K, Bhatt S, Luthra K. Effect of supervised progressive resistance-exercise training protocol on insulin sensitivity, glycemia, lipids, and body composition in Asian Indians with type 2 diabetes. Diabetes Care. 2008 Jul;31(7):1282-7. doi: 10.2337/dc07-2316. Epub 2008 Mar 3. PMID 18316394
- [Background] Maharaj, S. S., & Nuhu, J. M. (2015). The effect of rebound exercise and treadmill walking on the quality of life for patients with non-insulin-dependent type 2 diabetes. International Journal of Diabetes in Developing Countries, 35(October), 223-229. https://doi.org/10.1007/s13410-015-0350-z
- [Background] Beck AT, Steer RA, Ball R, Ranieri W. Comparison of Beck Depression Inventories -IA and -II in psychiatric outpatients. J Pers Assess. 1996 Dec;67(3):588-97. doi: 10.1207/s15327752jpa6703_13. PMID 8991972
- [Background] Arora E, Shenoy S, Sandhu JS. Effects of resistance training on metabolic profile of adults with type 2 diabetes. Indian J Med Res. 2009 May;129(5):515-9. PMID 19675378
- [Background] Cohen, J. (1977). Statistical power analysis for the behavioral sciences. Academic Press.
- [Background] Odole, A. C., & Akinpelu, A. O. (2009). Translation and Alternate Forms Reliability of the Visual Analogue Scale in the Three Major Nigerian Languages. Pain, 7(3), 1-7.
- [Background] Pai LW, Hung CT, Li SF, Chen LL, Chung Y, Liu HL. Musculoskeletal pain in people with and without type 2 diabetes in Taiwan: a population-based, retrospective cohort study. BMC Musculoskelet Disord. 2015 Nov 20;16:364. doi: 10.1186/s12891-015-0819-4. PMID 26589716
- [Background] International Diabetes Federation. (2013). IDF Diabetes Atlas. Hallado en: http://www. idf. org/diabetesatlas/5e/es/ …
- [Background] Who. (2001). The International Classification of Functioning, Disability and Health. World Health Organization, 18, 237. https://doi.org/10.1097/01.pep.0000245823.21888.71
- [Derived] Kaka B, Maharaj SS. Effect of Rebound Exercises and Circuit Training on Complications Associated with Type 2 Diabetes: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2018 May 7;7(5):e124. doi: 10.2196/resprot.8827. PMID 29735476